CLINICAL TRIAL: NCT06330480
Title: Check@Home: General Population Screening for Early Detection of Atrial Fibrillation and Chronic Kidney Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Folkert W. Asselbergs (Other)
Collaborators: Dutch Cardiovascular Alliance (Unknown); University Medical Center Groningen (Other); Dutch Heart Foundation (Other); Dutch Kidney Foundation (Other); Dutch Diabetes Research Foundation (Other); Maastricht University (Other); AstraZeneca (Industry); UMC Utrecht (Other); Radboud University Medical Center (Other); Siemens Healthineers Nederland BV (Unknown); University of Twente (Other); Roche Diagnostics Nederland BV (Unknown); Happitech BV (Unknown); Stichting Radboud Universiteit (Unknown); Stichting Netherlands Heart Institute (Unknown); Topicus.Healthcare BV (Unknown); Amsterdam UMC, location AMC (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Folkert W. Asselbergs, Prof. Dr. F. W. Asselbergs, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Check@Home
Record Dates: First submitted 2024-03-07; First posted 2024-03-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation; Chronic Kidney Diseases; Diabetes Mellitus, Type 2
Keywords: Population-based screening
MeSH Terms: conditions — Atrial Fibrillation; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Check@Home is a population-based screening with a phased assessment and implementation using an iterative design executed consecutively in four regions in the Netherlands.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Other): This group will be invited for the screening
  Interventions: Other: Intervention group
- Control group (No Intervention): This group will not be invited for the screening

INTERVENTIONS:
Other: Intervention group — Subjects will be invited for a home-based screening (phase 1) that includes home-based testing; urine collection for detection of elevated albuminuria, and a heart rhythm measurement for detection of atrial fibrillation. Both home-based tests will be performed with CE-marked medical devices used according to their intended use. A subset of the population will also receive a short questionnaire. Depending on the results of the home-based tests, subjects might be invited for further screening in a diagnostic screening facility (phase 2), that includes collection of physical data, blood, and urine for the assessment of parameters that are indicative of cardiovascular disease, chronic kidney disease, diabetes type 2 or their risk factors. Participants will also receive a questionnaire. Based on the results of the diagnostic screening, participants may be referred to their GP for appropriate treatment according to the prevailing guidelines (phase 3)
  Arms: Intervention group

SUMMARY:
The aim of the Check@Home consortium is to set up a roadmap and infrastructure for a program to early detect atrial fibrillation and chronic kidney disease in the general population.

This will be a population-based screening with a phased implementation and an iterative design in four regions in the Netherlands (Breda, Utrecht, Arnhem, Eindhoven). In total, a random sample of 160,000 people (aged 50-75 years) will be invited to participate in the study and another random sample of 160,000 people with the same characteristics will be included in the control group in which no screening will be offered.

The overall screening program will consist of three phases: a home-based testing phase, diagnostic screening phase, and a treatment phase:

* Phase 1: Subjects will be invited for a home-based screening that includes home-based testing; urine collection for detection of elevated albuminuria, and a heart rhythm measurement using a smartphone app for detection of atrial fibrillation.
* Phase 2: Depending on the results on these home-based tests, subjects will be invited for further screening in a diagnostic screening facility. During this visit, physical data will be collected (height, weight, waist circumference, blood pressure, heart rhythm), blood will be drawn, and urine will be collected for the assessment of parameters that are indicative of a cardiovascular disease, chronic kidney disease, type 2 diabetes or their risk factors. Participants will receive a questionnaire that include questions on demographics, educational level, disease history, medication use, health literacy, and quality of life.
* Phase 3: Based on the results of the diagnostic screening, participants may be referred to their general practitioner for appropriate treatment (lifestyle advice/medication) according to the prevailing guidelines.

The primary study outcomes are:

Overall effectiveness of population based screening on atrial fibrillation and chronic kidney disease in subjects aged 50-75 years, based on:

* Participation rate of different screening strategies and phases;
* Yield of the screening (number of subjects with (newly) diagnosed disease and risk factors);
* Effectiveness of the atrial fibrillation screening, compared with standard care, based on the incidence of ischemic stroke);
* Effectiveness of the albuminuria screening, compared with standard care, based on the incidence of kidney failure events and Major Adverse Cardiovascular Events (MACE).

DETAILED DESCRIPTION:
Background:

Currently, in the Netherlands there is no structured national approach for the early detection of cardiovascular disease, kidney disease, and type 2 diabetes in the general population, despite the social and economic impact of these disorders. Detecting these chronic conditions at an early stage could allow for adequate and early treatment to prevent the progression of these conditions and their complications, thereby reducing the societal and economic burden caused by these chronic diseases.

Objective of the study:

To investigate whether population-based screening of subjects aged 50-75 years can contribute to early detection and treatment of atrial fibrillation and chronic kidney disease (defined by elevated albuminuria), and thereby can contribute to prevention of the morbidity and mortality related to these diseases. This will be done by evaluating the participation rate, yield, and (cost-)effectiveness of the screening compared with standard care. Furthermore, the project aims to evaluate options for broader screening, including the early detection of heart failure, coronary artery disease, and type 2 diabetes.

Study design:

This will be a population-based screening with a phased implementation and an iterative design in four regions in the Netherlands (Breda, Utrecht, Arnhem, Eindhoven).

Participants will be invited for a home-based screening (phase 1) that includes home-based testing; urine collection for detection of elevated albuminuria as indicator of chronic kidney disease, and a heart rhythm measurement using a smartphone app for detection of atrial fibrillation. Both home-based tests will be performed with CE-marked medical devices used according to their intended use. A subset of the population will also receive a short questionnaire. Depending on the results of the home-based tests, subjects might be invited for further screening in a diagnostic screening facility (phase 2). During this visit, physical data (height, weight, waist circumference, blood pressure, heart rhythm) will be collected, blood will be drawn, and urine will be collected for the assessment of parameters that are indicative of a cardiovascular disease, chronic kidney disease, type 2 diabetes or their risk factors. Participants will receive a questionnaire that includes questions on demographics, educational level, disease history, medication use, health literacy, and quality of life. Based on the results of the diagnostic screening, participants may be referred to their general practitioner for appropriate treatment (lifestyle advice/medication) according to the prevailing guidelines. It is planned that in a future protocol amendment an alternative treatment trajectory will be added in which participants may receive further treatment in the diagnostic screening facility.

Study population:

In total, a random sample of 160,000 people (aged 50-75 years) living in one of the four selected regions in the Netherlands will be invited to participate in the study. Another random sample of 160,000 people (aged 50-75 years) living in one of the four selected regions in the Netherlands will be included in the control group in which no screening will be offered.

ELIGIBILITY:
Inclusion Criteria:

* aged between 50 and 75 years
* living in the selected regions (Breda, Utrecht, Arnhem, Eindhoven)

Exclusion Criteria:

* age <50 years or >75 years
* not living in the selected regions (Breda, Utrecht, Arnhem, Eindhoven)
* being institutionalized (e.g., subjects with intellectual disabilities or subjects living in nursing homes who have a limited life expectancy)
* participants of the previously conducted THOMAS Study (NL65228.042.18, METc 2018/687) will be excluded.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320000 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Participation rate of the atrial fibrillation and albuminuria screening | 1 year after screening period
  * Participation rate of the home-based screening phase will be defined as the number of persons who completed the home-based screening phase relative to the number of persons invited in the corresponding arm (intention-to-screen);
  * Participation rate of the diagnostic screening phase will be defined as the number of persons who completed the diagnostic screening phase relative to the number of persons invited for the diagnostic screening phase in the corresponding arm (in participants invited based on an 'abnormal' result in the home-based screening phase, i.e. either confirmed elevated albuminuria or an irregular heart rhythm);
  * Participation rate of the treatment phase will be defined as the number of persons who completed the care initiation phase (i.e., number of participants visiting their GP; or - in future phases of the screening - the diagnostic center) relative to the number of persons referred for treatment in the corresponding arm (intention-to-screen).
Yield of the atrial fibrillation and albuminuria screening | 1 year after screening period
  * Yield of home-based screening: number of participants tested positive (i.e., either confirmed positive urine test and/or abnormal heart rhythm test) relative to the number of persons participating in the corresponding arm (per-protocol analysis) and to the number of persons invited in the corresponding arm (intention-to-screen analysis);
  * Yield of diagnostic screening: number of participants with (newly) diagnosed cardiovascular or chronic kidney disease, diabetes or risk factors, relative to the number of persons participating in the corresponding arm (per-protocol analysis) and to the number of persons invited in the corresponding arm (intention-to-screen analysis);
  * Yield of treatment phase: number of participants completing the treatment phase relative to the number of persons participating in the corresponding arm (per-protocol analysis) and to the number of persons invited to the treatment phase in the corresponding arm (intention-to-screen analysis).
Effectiveness of the atrial fibrillation screening | Up to 10 years follow-up after screening period
  Effectiveness of the atrial fibrillation screening (the home-based screening program and follow-up strategy) will be based on the incidence of (fatal and non-fatal) ischemic stroke. This will be evaluated by comparing the event rates in the intervention group (the sample of 160,000 subjects invited for screening) and the control group (the sample of 160,000 subjects not invited for screening).
Effectiveness of the albuminuria screening | Up to 10 years follow-up after screening period
  Effectiveness of the albuminuria screening (the home-based screening program and follow-up strategy), based on the incidence of the composite outcome of kidney failure events (defined as start of dialysis, receiving a kidney transplant, or death due to kidney failure without having started kidney function replacement treatment) and MACE (for albuminuria screening defined as cardiovascular mortality, stroke, and myocardial infarction, including CABG and PCI).
  This will be evaluated by comparing the event rates in the population screened positive for elevated albuminuria and followed-up based on this result (i.e., participants in the standard strategy and other alternative strategies) and in the population screened positive for elevated albuminuria - at a later timepoint - and not followed-up based on this result (i.e., participants in 'alternative strategy B').

SECONDARY OUTCOMES:
Effectiveness of the atrial fibrillation screening based on incidence of MACE events | Up to 10 years follow-up after screening period
  Effectiveness of the atrial fibrillation screening (the home-based screening program and follow-up strategy), based on the incidence of MACE (for atrial fibrillation screening defined as cardiovascular mortality, stroke, non-hemorrhagic stroke, and myocardial infarction, including CABG and PCI).
  This will be evaluated by comparing the event rates in the intervention group (the sample of 160,000 subjects invited for screening) and the control group (the sample of 160,000 subjects not invited for screening).
Effectiveness of the albuminuria screening based on incidence each individual MACE component | Up to 10 years follow-up after screening period
  Effectiveness of the albuminuria screening (the home-based screening program and follow-up strategy), based on each individual component defining MACE (for albuminuria screening defined as cardiovascular mortality, stroke, and myocardial infarction, including CABG and PCI).
  This will be evaluated by comparing the event rates in the in the population screened positive for elevated albuminuria and followed-up based on this result (i.e., participants in the standard strategy and other alternative strategies) and in the population screened positive for elevated albuminuria - at a later timepoint - and not followed-up based on this result (i.e., participants in 'alternative strategy B').
Safety of the atrial fibrillation screening | Up to 10 years follow-up after screening period
  Safety of the atrial fibrillation screening (the home-based screening program and follow-up strategy), based on the incidence of the composite outcome of (fatal and non-fatal) hemorrhagic stroke, other major bleeding events leading to hospitalization (including but not limited to intracranial bleeds, sight-threatening eye bleeds, and serious gastrointestinal bleeding), and all cause-mortality.
  This will be evaluated by comparing the event rates in the intervention group (the sample of 160,000 subjects invited for screening) and the control group (the sample of 160,000 subjects not invited for screening).
Cost-effectiveness of screening strategies compared with standard of care: treatment effectiveness based on literature. | Up to 10 years follow-up after screening period
  An individual level simulation model will be developed to estimate the lifetime effects of the screening strategies for the detection of atrial fibrillation and chronic kidney disease by comparing the corresponding expected incidences of cardiovascular and chronic kidney disease, diabetes and their complications and endpoints with standard care. Incremental effectiveness will be calculated, expressed in QALYs gained for the different screening strategies. Costs will be calculated by multiplying resource use with the corresponding unit costs. The ICER between screening strategies and no screening, expressed in costs per QALY gained, will be calculated over a short-time (5-10 years after screening) and a lifetime time horizon. Finally, we will assess the chance that screening is cost-effective for a range of willingness-to-pay threshold values (range €20,000-€80,000 per QALY) and at which threshold for the screening costs screening would have a chance of ≥90% to be cost-effective.
Cost-effectiveness of screening strategies compared to standard of care: treatment effectiveness based on actual observed event rates | Up to 10 years follow-up after screening period
  Using registry data, we will compare event rates between the intervention group (invited for screening) and the control group (not invited for screening) 5 and 10 years after the screening. Currently foreseen is that the data on fatal and non-fatal cardiovascular disease (according to the MACE criteria; based on corresponding ICD-10 codes) and renal events (dialysis and transplantation; based on corresponding ICD-10 codes) will be obtained and compared. These data will be obtained by linkage with CBS (i.e., Dutch Hospital Data, Vektis, Zorginstituut Nederland), Zorgverzekeraars Nederland, Pharmo, National Heart Registry, and general practitioner registries. These data will be input for the health economic simulation model, replacing earlier estimates of treatment effectiveness and treatment adherence. The ICER and estimation of the likelihood of screening being cost-effective will be repeated using this new and more accurate evidence.

OTHER OUTCOMES:
False-positive rate, false-negative rate, sensitivity, specificity, positive predictive screening on atrial fibrillation and albuminuria screening. | Up to 10 years follow-up after screening period
  * False-positives: participants with an abnormal home-based test result, but normal test results at the diagnostic screening visit.
  * False-negatives: participants with normal home-based test results, but abnormal test results at the diagnostic screening visit.
  * Sensitivity: the ability of the home-based test to correctly identify participants with the disease.
  * Specificity: the ability of the home-based test to correctly identify participants without the disease.
  * Positive predictive value: the proportion of participants correctly diagnosed as positive (having the disease) out of all participants with a positive test result.
  * Negative predictive value: the proportion of participants correctly diagnosed as negative (not having the disease) out of all participants with a negative test result.
Characteristics of responders and non-responders | Up to 10 years follow-up after screening period
  Characteristics of responders and non-responders, and differences between them, will be analyzed using descriptive statistics per screening strategy. For health literacy descriptive statistical analyses will be performed on the HLS-Q12 questionnaire (per item and/or combined). Future exploratory analyses may evaluate whether health literacy is related to participation rate, health outcomes, and or characteristics of participants and non-participants (such as age and socioeconomic indicators of the neighborhood). In addition, facilitators and barriers for participation will be studied taking into account qualitative data on experiences, considerations and enabling and constraining conditions, collected both in participants and non-participants via in-depth interviews and/or observations.
Effectiveness of the atrial fibrillation screening based on incidence each individual MACE component | Up to 10 years follow-up after screening period
  Effectiveness of the atrial fibrillation screening (the home-based screening program and follow-up strategy), based on the incidence of each individual component defining MACE (for the atrial fibrillation screening defined as cardiovascular mortality, non-hemorrhagic stroke, and myocardial infarction, including CABG and PCI).
  This will be evaluated by comparing the event rates in the intervention group (the sample of 160,000 subjects invited for screening) and the control group (the sample of 160,000 subjects not invited for screening).
Overall effectiveness of broader population-based screening strategies applied to screening on heart failure, coronary artery disease, and type 2 diabetes. | Up to 10 years follow-up after screening period
  Overall effectiveness of broader population-based screening strategies, focused on the detection (and potentially treatment) of heart failure, coronary artery disease, and type 2 diabetes in subjects aged 50-75 years. This will be evaluated based on participation rate, yield, and (cost-)effectiveness of the screening strategies, similarly to what is described in the previous sections, but then applied to screening on heart failure, coronary artery disease, and type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. F. W. Asselbergs, Principal Investigator — Amsterdam UMC; Prof. Dr. R. T. Gansevoort, Principal Investigator — UMC Groningen
Locations (1):
- Stichting Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Mil D, Kieneker LM, Evers-Roeten B, Thelen MHM, de Vries H, Hemmelder MH, Dorgelo A, van Etten RW, Heerspink HJL, Gansevoort RT. Participation rate and yield of two home-based screening methods to detect increased albuminuria in the general population in the Netherlands (THOMAS): a prospective, randomised, open-label implementation study. Lancet. 2023 Sep 23;402(10407):1052-1064. doi: 10.1016/S0140-6736(23)00876-0. Epub 2023 Aug 16. PMID 37597522
- See also: Related Info — https://checkathome.nl